CLINICAL TRIAL: NCT00775593
Title: An Open Label Phase II Trial of Clofarabine and Temsirolimus in Older Patients With Relapsed or Refractory Acute Myeloid Leukemia (AML)
Brief Title: Clofarabine and Temsirolimus in Treating Older Patients With Relapsed or Refractory Acute Myeloid Leukemia
Acronym: AML1107
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML1107; GIMEMA-AML-1107; EUDRACT-2007-005374-31
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with inv(16)(p13;q22)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myelomonocytic, Acute; Congenital Abnormalities | interventions — Clofarabine; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: clofarabine — Patients will receive one course of low-dose Clofarabine in combination with Temsirolimus (CloTor regimen) for remission induction.
  Induction therapy
  - Clofarabine 20 mg/m2/day, administered by iv infusion over 1 hour on days 1 through 5
Drug: temsirolimus — Those who achieve morphologic CR and morphologic CRi will receive maintenance treatment with Temsirolimus monthly for 12 months, or until relapse.
  Those who achieve a PR will receive one additional course of CloTor and, if a CR/CRi is obtained, maintenance treatment with Temsirolimus as above.
  Induction therapy:
  - Temsirolimus 25 mg (flat dose) administered iv over 30 minutes on days 1, 8 and 15.
  Maintenance therapy:
  - Temsirolimus 25 mg (flat dose) administered iv over 30 minutes on days 1 and 8 of each month for 12 months, or until relapse.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as clofarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Temsirolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving clofarabine together with temsirolimus may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving clofarabine together with temsirolimus works in treating older patients with relapsed or refractory acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the complete response rate in older patients with relapsed or refractory acute myeloid leukemia when treated with low-dose clofarabine and temsirolimus.

Secondary

* To determine the tolerability and safety of this regimen.
* To determine the duration of response.
* To determine the duration of survival.

OUTLINE: This is a multicenter study.

* Induction therapy: Patients receive clofarabine IV over 1 hour on days 1-5 and temsirolimus IV over 30 minutes on days 1, 8, and 15. Treatment continues for 1-2 courses in the absence of disease progression or unacceptable toxicity.
* Maintenance therapy: Patients achieving morphologic complete remission (CR) or CR with incomplete blood count recovery receive temsirolimus IV over 30 minutes on days 1 and 8 of each month. Treatment continues for 12 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically confirmed acute myeloid leukemia (AML) meeting the following criteria:

  * At least 20% of blasts in the bone marrow
  * AML in first relapse OR refractory to no more than one prior combination of intensive chemotherapy induction regimen
* No acute promyelocytic leukemia
* No blast transformation of chronic myeloid leukemia or other myeloproliferative disorders
* No active CNS leukemia

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Life expectancy ≥ 4 weeks
* Serum total bilirubin ≤ 1.5 times upper limit of normal (ULN)*
* AST and ALT ≤ 2.5 times ULN*
* Serum creatinine ≤ 1.0 mg/dL* OR estimated glomerular filtration rate > 60 mL/min
* No active uncontrolled systemic infection
* No concurrent active malignancy
* No HIV positivity
* No severe concurrent medical condition or psychiatric disorder that would preclude study participation NOTE: *Unless due to organ leukemic involvement

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior myelosuppressive chemotherapy
* At least 48 hours since prior hydroxyurea
* No prior clofarabine or temsirolimus
* No prior allogeneic stem cell transplantation
* No investigational drug within the past 30 days

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-12; Primary Completion 2012-06 (Actual); Study Completion 2013-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Amadori, MD, Principal Investigator — Ospedale Sant' Eugenio
Locations (19):
- Italy (19):
  - Azienda ospedaliera Nuovo ospedale "Torrette", Ancona
  - Azienda Ospedaliero-Universitaria Policlinico Consorziale, Bari
  - Azienda Ospedaliera Di Bologna Policlinico S. Orsola - Malpighi, Bologna
  - Ospedale Ferrarotto, Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Azienda ospedaliera di Rilievo Nazionale "A. Cardarelli", Napoli
  - Azienda Ospedaliera Universitaria - Università degli Studi di Napoli "Federico II" - Facoltà di Medicina e Chirurgia, Napoli
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - A.O. Universitaria S. Luigi Gonzaga di Orbassano, Orbassano
  - Azienda Ospedaliero - Universitaria di Parma, Parma
  - Azienda ASL di Pescara, Pescara
  - Complesso Ospedaliero S. Giovanni Addolorata, Roma
  - Ospedale S. Eugenio, Roma
  - S.C. di Ematologia e Trapianti - I.F.O. Istituto Nazionale Tumori Regina Elena, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Policlinico di Tor Vergata, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Serv. di Ematologia Ist. di Ematologia ed Endocrinologia, Sassari
  - Policlinico G. B. Rossi - Borgo Roma, Verona

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between April 2009 and June 2010, 60 patients were enrolled in the study at 14 different Italian institutions.
Groups:
- Study Group: Patients will receive one course of low-dose Clofarabine in combination with Temsirolimus (CloTor regimen) for remission induction. Those who achieve morphologic complete remission (CR) and morphologic complete remission with incomplete blood count recovery (CRi) will receive maintenance treatment with Temsirolimus monthly for 12 months, or until relapse. Those who achieve a partial remission (PR) will receive one additional course of CloTor and, if a CR/CRi is obtained, maintenance treatment with Temsirolimus as above. Patients not achieving CR or CRi after one or two induction courses will be discontinued from the study.
Period: Overall Study
Arm/Group | Study Group
Started | 60
Completed | 53
Not Completed | 7
Not completed — Unmet eligibility criteria | 6
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 53
Age, Customized [Mean (Full Range); unit: Years] | 69 [60 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 31
Region of Enrollment [Number; unit: participants]
  Italy | 53

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate
Time Frame: At 2 years from study entry
Measure: Number; unit: participants
Groups:
- Study Group: Evaluable patients
Arm/Group | Study Group
Number analyzed (Participants) | 53
participants | 4

2. Secondary Outcome: Number of Serious Adverse Events Within 2 Years
Time Frame: At 2 years from study entry
Measure: Number; unit: serious adverse events
Arm/Group | Study Group
Number analyzed (Participants) | 53
serious adverse events | 22

3. Secondary Outcome: Duration of Response
Description: Participants who responded to treatment
Time Frame: At 2 years from study entry
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Study Group
Number analyzed (Participants) | 11
months | 3.5 (12)

4. Secondary Outcome: Duration of Survival
Time Frame: At 2 years from study entry
Measure: Median (Full Range); unit: months
Arm/Group | Study Group
Number analyzed (Participants) | 53
months | 10.9 [0.3 to 20.2]

ADVERSE EVENTS:
Description: Non-serious adverse events have not been analyzed
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 15/53
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=53)
Cardiac arrest (Cardiac disorders) | 1 (1)
Gastrointestinal mucositis (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Disease Progression (General disorders) | 4 (4)
Mucosal inflammation (General disorders) | 1 (1)
E. coli sepsis (Infections and infestations) | 1 (1)
Pseudomonal sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Cerebral ischemia (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1)
Optic ischaemic neuropathy (Nervous system disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results are analyzed together with the sponsor, being the present study a fully independent not-for-profit trial.